CLINICAL TRIAL: NCT02733276
Title: Randomized Study : Electroacupuncture vs. Sham Electroacupuncture for Treatment of Fatigue in Patients With Inflammatory Bowel Disease
Brief Title: Electroacupuncture vs. Sham Electroacupuncture for Treatment of Fatigue in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana Horta-Sangenis, Resident Physician, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014067
Record Dates: First submitted 2016-03-05; First posted 2016-04-11 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Fatigue; Inflammatory Bowel Disease
MeSH Terms: conditions — Fatigue; Inflammatory Bowel Diseases | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Electroacupuncture (Experimental): Using electroacupuntor with different frequencies during 20 minutes. Needles are connected to the electrodes. Acupoints are: 6 needles in each lower limb, 8 abdominal, 3 in upper extremity and 3 on the front
  Interventions: Other: electroacupuncture
- Electroacupuncture sham (Sham Comparator): Using electroacupuntor with different frequencies during 20 minutes. Needles are connected to the electrodes. Acupoints are: needles on each forearm on nonselective points
  Interventions: Other: Sham: Electroacupuncture sham
- Control (No Intervention): Initially no intervention. In a second period in this group we will perform EAP

INTERVENTIONS:
Other: electroacupuncture — Electroacupuncture: Using an electroacupuntor with different frequencies during 20 minutes. Needles are connected to the electrodes.
  Arms: Electroacupuncture
Other: Sham: Electroacupuncture sham — Sham comparator (Electroacupuncture sham): Using an electroacupuntor with different frequencies during 20 minutes. Needles are connected to the electrodes.
  Arms: Electroacupuncture sham

SUMMARY:
Fatigue is a common symptom in inflammatory bowel diseaseI and persists despite clinical remission. Fatigue in patients with chronic diseases can be objectified by the FACIT-F scale. Acupuncture has been shown useful in the treatment of fatigue in various chronic diseases.

This study evaluates the effect of electroacupuncture in the treatment of fatigue in patients with quiescent inflammatory bowel disease.

Patients with inflammatory bowel disease and severe fatigue (FACIT-F score <38) who agree to participate in the study will be randomized to three different treatments: electroacupuncture vs. sham electroacupuncture vs. control group.

DETAILED DESCRIPTION:
Fatigue is a common symptom in inflammatory bowel disease and persists despite clinical remission. Fatigue in patients with chronic diseases can be objectified by the FACIT-F scale. Acupuncture has been shown useful in the treatment of fatigue in various chronic diseases.

This study evaluates the effect of electroacupuncture in the treatment of fatigue in patients with quiescent inflammatory bowel disease.

Patients with inflammatory bowel disease and severe fatigue (FACIT-F score < 38) who agree to participate in the study will be randomized to three different treatments: electroacupuncture vs. sham electroacupuncture vs. group control.

Treatment consists of a total of 9 sessions / patient (2 sessions / week the first week and then one session / week for two months).

During and after treatment, patients fill in questionnaires to assess fatigue, anxiety, depression, quality of life in inflammatory bowel disease and sleepiness. Those patients who do not improve with the initial treatment or present a recurrence of fatigue (defined as a decrease of at least 4 points in the FACIT-F score) then receive crossover treatment for 8 more weeks (total of 9 new sessions).

The control group fill in questionnaires in the same periods as patients who receive active treatment. These patients (control group) receive electroacupuncture sessions(total of 9 sessions) in a second period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease and fatigue in patients over 18 years
* Presence of continued fatigue determined in two consecutive scores and stability of the symptoms of fatigue according to the patient's opinion .
* Inflammatory bowel disease diagnosed at least 6 months before the study (diagnosed by clinical, laboratory , endoscopic and histological criteria) .
* Written informed consent

Exclusion Criteria:

* Patients who are participating in other clinical studies.
* Associated tumor disease .
* Pregnant or breast feeding women .
* Anemia Hemoglobin determined under 12 in women and 14 in men.
* Patients who have suffered minor adverse reactions to acupuncture.
* Prior Acupuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of acupuncture in the treatment of fatigue in patients with inflammatory bowel disease (assessed by the FACIT-F scale). | 7 months
  Assessed by the FACIT-F scale

SECONDARY OUTCOMES:
Evaluate the effectiveness of acupuncture in the treatment of depression in patients with fatigue and inflammatory bowel disease (assessed by the Depression Beck scale). | 7 months
  assessed by the Depression Beck scale
Evaluate the effectiveness of acupuncture in the treatment of anxiety in patients with fatigue and inflammatory bowel disease (assessed by the Hamilton scale). | 7 months
  assessed by the Hamilton scale
Evaluate the effectiveness of acupuncture in the treatment of sleepiness in patients with fatigue and inflammatory bowel disease (assessed by the Epworth scale). | 7 months
  assessed by the Epworth scale

CONTACTS AND LOCATIONS:
Overall Officials: Diana Horta, Principal Investigator — Parc Tauli Hospital
Locations (1):
- Diana Horta, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horta D, Lira A, Sanchez-Lloansi M, Villoria A, Teggiachi M, Garcia-Rojo D, Garcia-Molina S, Figuerola A, Esteve M, Calvet X. A Prospective Pilot Randomized Study: Electroacupuncture vs. Sham Procedure for the Treatment of Fatigue in Patients With Quiescent Inflammatory Bowel Disease. Inflamm Bowel Dis. 2020 Feb 11;26(3):484-492. doi: 10.1093/ibd/izz091. PMID 31091322